CLINICAL TRIAL: NCT07105514
Title: Indole-3-PROpionic Acid Clinical Trials - a Pilot Study Part 2 (iPROACT-pilot2)
Brief Title: Indole-3-PROpionic Acid Clinical Trials - a Pilot Study Part 2
Acronym: iPROACT-pilot2
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Glostrup University Hospital, Copenhagen (Other)
Collaborators: University of Copenhagen (Other); University of Southampton (Other)
Responsible Party: Principal Investigator, Jette Lautrup Frederiksen, Prof, DMSc, MD, Glostrup University Hospital, Copenhagen
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: H-24008127 - 116180
Record Dates: First submitted 2025-07-17; First posted 2025-08-06 (Actual); Last update posted 2025-08-08 (Actual); Status verified 2025-08

CONDITIONS: Healthy
Keywords: indole-3-propionic acid; gut bacterial metabolite; regulatory T cells; brain-derived neurotrophic factor; dietary supplement

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Randomization is performed by external party. Each capsule container is labelled with a unique number (101-160) and no other identifier. Capsule containers have already been randomized by the external party using block randomization with random block sizes of 2 or 4. Study participants receive the next available capsule container based on their order of recruitment. This way, everyone involved in the study is fully blinded and it is also impossible to guess which participants belong to the same group. Only after all study participants have been recruited and the collected data have been cleaned and quality checked, are the researchers performing the statistical analyses informed about which participants belong to the same group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator): Placebo
  Interventions: Dietary Supplement: Placebo
- Indole-3-propionic acid (IPA) (Experimental): IPA: total daily dose of 1000 mg
  Interventions: Dietary Supplement: Indole-3-propionic acid (IPA)

INTERVENTIONS:
Dietary Supplement: Indole-3-propionic acid (IPA) — Two capsules are taken every morning and two capsules are taken every evening for 14 consecutive days. Active capsules are taken orally and contain 250 mg of IPA each.
  Arms: Indole-3-propionic acid (IPA)
Dietary Supplement: Placebo — Two capsules are taken every morning and two capsules are taken every evening for 14 consecutive days. Placebo capsules are taken orally and contain maltodextrin.
  Arms: Placebo

SUMMARY:
The goal of this trial is to investigate the biological effects of oral supplementation with indole-3-propionic acid (IPA) taken twice daily in healthy adults. The main scientific questions are:

* Does supplementation with IPA increase the abundance of regulatory T cells in the blood? Regulatory T cells are believed to play an important role in preventing autoimmune diseases.
* Does supplementation with IPA increase the concentration of brain-derived neurotrophic factor (BDNF) in the blood? BDNF is believed to play an important role in maintaining brain health.
* Does supplementation with IPA affect blood analyses commonly performed to assess the risk of metabolic disorders like type 2 diabetes and cardiovascular diseases?

Participants will:

* Take capsules to achieve a total daily dose of 1000 mg of IPA or placebo: 500 mg every morning and 500 mg every evening for 14 days.
* Visit the clinic at the beginning (day 1) and at the end (day 15) of the supplementation period to deliver blood, urine and fecal samples, have simple measurements performed, fulfil questionnaires and report any side effects.

DETAILED DESCRIPTION:
Indole-3-propionic acid (IPA) is a gut bacterial metabolite with the amino acid tryptophan as substrate. In vitro and animal studies suggest that IPA could contribute to regulating inflammation and metabolic function, preventing oxidative damage and upregulating expression of brain-derived neurotrophic factor. With this study we aim to investigate the biochemical effects of IPA at supraphysiological levels in humans.

ELIGIBILITY:
Inclusion Criteria:

* Healthy women and men ≥18 and ≤65 years of age
* Deemed mentally and physically able to participate

Exclusion Criteria:

* Diagnosis of gut-, heart-, liver-, kidney or immune-related disorders
* Use of antibiotics within the last month
* Pregnancy, lactation or childbirth within the last five months
* Use of prescription medication

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2025-08-04 (Actual); Primary Completion 2025-10-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Regulatory T cells (first primary outcome) | Results from fasting blood samples taken on day 15 and adjusted for results from day 1 (fasting just before first supplement/placebo dose).
  FoxP3+CD25+CD127- regulatory T cells expressed as a percentage of single, live CD3+CD4+CD8- lymphocytes. Analysed in freshly isolated peripheral blood mononuclear cells using a Symphony A3 flowcytometer.
Brain-derived neurotrophic factor (second primary outcome) | Results from fasting blood samples taken on day 15 and adjusted for results from day 1 (fasting just before first supplement/placebo dose).
  Brain-derived neurotrophic factor measured in platelet-free plasma samples using ELISA or mesoscale.

SECONDARY OUTCOMES:
Th1/Th2 ratio in PBMCs | Results from fasting blood samples taken on day 15 and adjusted for results from day 1 (fasting just before first supplement/placebo dose).
  Th1/Th2 ratio calculated from T cell profiling of freshly isolated peripheral blood mononuclear cells (PBMCs) using a Symphony A3 flowcytometer.
  Th1 cells are defined as the CXCR3+CCR4-CCR6-CCR10- non-Treg population and expressed as a percentage of single, live CD3+CD4+CD8-CD45RA- lymphocytes.
  Th2 cells are defined as the CXCR3-CCR4+CCR6-CCR10- non-Treg population and expressed as a percentage of single, live CD3+CD4+CD8-CD45RA- lymphocytes.
  Panel antigens: FVS780, CD3, CD4, CD8, CD45RA, CCR7, CXCR3, CCR6, CCR4, CCR10, CD25, CD127, FoxP3.
Th17/mTreg ratio in PBMCs | Results from fasting blood samples taken on day 15 and adjusted for results from day 1 (fasting just before first supplement/placebo dose).
  Th17/mTreg ratio calculated from T cell profiling of freshly isolated peripheral blood mononuclear cells (PBMCs) using a Symphony A3 flowcytometer.
  Th17 cells are defined as the CXCR3-CCR4+CCR6+CCR10- non-Treg population and expressed as a percentage of single, live CD3+CD4+CD8-CD45RA- lymphocytes.
  mTreg (memory Tregs) are defined as the FoxP3+CD25+CD127-CD45RA- population and expressed as a percentage of single, live CD3+CD4+CD8-CD45RA- lymphocytes
  Panel antigens: FVS780, CD3, CD4, CD8, CD45RA, CCR7, CXCR3, CCR6, CCR4, CCR10, CD25, CD127, FoxP3.
Th17.1 cells in PBMCs | Results from fasting blood samples taken on day 15 and adjusted for results from day 1 (fasting just before first supplement/placebo dose).
  Th17.1 cells in freshly isolated peripheral blood mononuclear cells (PBMCs) characterized using a Symphony A3 flowcytometer.
  Th17.1 cells are defined as the CXCR3+CCR4-CCR6+CCR10- non-Treg population and expressed as a percentage of single, live CD3+CD4+CD8-CD45RA- lymphocytes
  Panel antigens: FVS780, CD3, CD4, CD8, CD45RA, CCR7, CXCR3, CCR6, CCR4, CCR10, CD25, CD127, FoxP3.
CRP | Results from blood samples taken on day 15 (just before last supplement/placebo dose) and adjusted for results from day 1 (just before first supplement/placebo dose).
  C-reactive protein (CRP) measured in plasma (mg/L) as a biomarker of infection and systemic inflammation. Lower-limit of quantification: 0,4 mg/L. Values below 0,4 mg/L are imputed as 0,2 mg/L.
Triglycerides | Results from fasting blood samples taken on day 15 and adjusted for results from day 1 (fasting just before first supplement/placebo dose).
  Plasma triglycerides (mmol/l).
non-HDL cholesterol | Results from fasting blood samples taken on day 15 and adjusted for results from day 1 (fasting just before first supplement/placebo dose).
  Non-HDL cholesterol calculated as total cholesterol minus HDL cholesterol (mmol/l)
C-peptide | Results from fasting blood samples taken on day 15 and adjusted for results from day 1 (fasting just before first supplement/placebo dose).
  Proinsulin C-peptide (pmol/l) measured in plasma.
Fasting glucose | Results from fasting blood samples taken on day 15 and adjusted for results from day 1 (fasting just before first supplement/placebo dose).
  Plasma glucose (mmol/l). Participants abstain from eating and drinking after 22.00 the day before. Only water is allowed. Fasting blood samples are taken between 8.00-10.00 in the morning.
F2-isoprostanes | Results from samples taken on day 15 and adjusted for results from day 1.
  F2-isoprostanes with a specific focus on 8-iso-prostaglandin F2α measured in blood or morningurine samples as a marker of lipid oxidation.
8-oxo-dG | Results from samples taken on day 15 and adjusted for results from day 1.
  8-oxo-dG (8-Oxo-2'-deoxyguanosine) measured in blood or morningurine samples as a marker of DNA-related stress damage.
Serum metabolomics | Four samples in total. Day 1 prior to and again 1.5 hour after intake of first capsule of IPA/ placeblo. Day 15 prior to and again 1.5 hour after intake of last capsule of IPA/ placebo.
  Targetted and untargetted liquid-chromatography mass-spectrometry-based metabolomics of serum samples. Targetted analyses aim to quantify indole-3-propionic acid and its metabolites (biomarker of compliance as well as absorptive and metabolic capacity), other bacterial- and host metabolites of tryptophan as well as short-chain fatty acids.
Total cholesterol | Results from fasting blood samples taken on day 15 and adjusted for results from day 1 (fasting just before first supplement/placebo dose).
  Plasma cholesterol (mmol/l).
VLDL cholesterol | Results from fasting blood samples taken on day 15 and adjusted for results from day 1 (fasting just before first supplement/placebo dose).
  Plasma very low-density lipoproteins (mmol/l).
LDL cholesterol | Results from fasting blood samples taken on day 15 and adjusted for results from day 1 (fasting just before first supplement/placebo dose).
  Plasma low-density lipoprotein (LDL) (mmol/l).
HDL cholesterol | Results from fasting blood samples taken on day 15 and adjusted for results from day 1 (fasting just before first supplement/placebo dose).
  Plasma high-density lipoprotein (HDL) (mmol/l).
Malondialdehyde | Results from samples taken on day 15 and adjusted for results from day 1.
  Malondialdehyde measured in blood or morningurine samples as a marker of oxidative stress.
Protein carbonyls | Results from samples taken on day 15 and adjusted for results from day 1.
  Protein carbonyls measured in blood or morningurine samples as a marker of protein oxidation.
Glycated hemoglobin (HbA1c) | Results from fasting blood samples taken on day 15 and adjusted for results from day 1 (fasting just before first supplement/placebo dose).
  HbA1c (IFCC, mmol/mol) measured in whole blood. Estimated average glucose values (mmol/l) are also calculated automatically from HbA1c by our laboratory.
T cell profiling | Results from fasting blood samples taken on day 15 and adjusted for results from day 1 (fasting just before first supplement/placebo dose).
  Targetted and untargetted T cell profiling of freshly isolated peripheral blood mononuclear cells (PBMCs) using a Symphony A3 flowcytometer. Panel antigens: FVS780, CD3, CD4, CD8, CD45RA, CCR7, CXCR3, CCR6, CCR4, CCR10, CD25, CD127, FoxP3.
  Target populations:
  Naïve: CD45RA+CCR7+, Central memory: CD45RA-CCR7+, Effector memory: CD45RA-CCR7-, TEMRA: CD45RA+CCR7-, Th1: CXCR3+CCR4-CCR6-CCR10-, Th2: CXCR3-CCR4+CCR6-CCR10-, Th17: CXCR3-CCR4+CCR6+CCR10-, Th17.1: CXCR3+CCR4-CCR6+CCR10-, Th22: CXCR3-CCR4+CCR6+CCR10+, as well as expression of chemokine receptors on cytotoxic T cells and regulatory T cells.
  An untargetted approach may be employed to allow for unbiased identification of changes in novel, yet uncharacterized populations.
Changes in the gut microbiome | Fecal samples are collected at three time points: prior to supplementation (earliest 48 hours prior to first visit (day 1)), short after initiation of supplementation (day 3 or soonest thereafter) and again earliest 48 hours prior to last visit.
  Characterization of the gut microbiome using molecular biology methods such as 16s rRNA sequencing.
Characterization of the metabolic activity of the gut microbiota | Fecal samples are collected at three time points: prior to supplementation (earliest 48 hours prior to first visit (day 1)), short after initiation of supplementation (day 3 or soonest thereafter) and again earliest 48 hours prior to last visit.
  Targetted and untargetted liquid-chromatography mass-spectrometry-based metabolomics. Targetted analyses aim to quantify indole-3-propionic acid, other bacterial- and host metabolites of tryptophan as well as short-chain fatty acids.
Bacterial polysaccharides | Results from samples taken on day 15 and adjusted for results from day 1.
  Endotoxin, capsular polysaccharides or other bacterial polysaccharides measured in blood samples as biomarker of bacterial translocation across the intestinal epithelium.
Pre-haptoglobin 2 | Results from samples taken on day 15 and adjusted for results from day 1.
  Measurement of pre-haptoglobin 2 in blood samples as a biomarker of intestinal permeability.
Intestinal fatty acid binding protein | Results from samples taken on day 15 and adjusted for results from day 1.
  Measurements of intestinal fatty acid binding protein in blood samples as a biomarker of enterocyte damage.
Citrulline | Results from samples taken on day 15 and adjusted for results from day 1.
  Measurement of citrulline in blood samples as a biomarker of intestinal function.
Calprotectin | Results from samples taken on day 15 and adjusted for results from day 1.
  Calprotectin measured in fecal samples as a biomarker of intestinal inflammation.
Neopterin | Results from samples taken on day 15 and adjusted for results from day 1.
  Neopterin measured in morningurine samples as a biomarker of systemic inflammation.
suPAR | Results from samples taken on day 15 and adjusted for results from day 1.
  Soluble urokinase plasminogen activator receptor (suPAR) measured in blood samples.
Microvesicles | Results from samples taken on day 15 and adjusted for results from day 1.
  Flow cytometric analyses of microvesicles/ microparticles in platelet-free plasma as biomarker of systemic inflammation.
Endothelial progenitor cells | Results from samples taken on day 15 and adjusted for results from day 1.
  Flow cytometric analyses of endothelial progenitor cells measured in platelet-free plasma as biomarker of systemic inflammation

OTHER OUTCOMES:
Gastrointestinal comfort | Gastrointestinal symptoms are assessed on day 1 and day 15.
  Self-reported (questionnaire) gastrointestinal symptoms of bloating, pain, rumbling, flatulence, constipation, hard stools and diarrhea evaluated using a visual analogue scale as well as a question on the frequency of defecation.
Gastrointestinal transit time | The maize test is performed at baseline (maize is ingested five days before visit 1) and repeated on day 10 (five days before visit 2).
  Measurement of transit time through the digestive system using a so-called maize test. Participants consume 100 grams of sweet maize in the morning between 5.30-10.00 while still in a fasting state. The exact date and time of consumption is registered and so is the exact date and time when maize is observed for the first time in feces. Transit time is expressed as the difference between the ingestion and fecal excretion timepoints in hours.
Stool consistency | Bristol stool chart is used in association with each maize test and collection of fecal samples (earliest 48 hours prior to first visit and day 3 or soonest thereafter and again earliest 48 hours prior to last visit (day 15)).
  Classification of stool consistency using the Bristol Stool Chart. Numerical scale ranging from 1 (separate hard lumps) to 7 (liquid consistency with no solid pieces) with one-unit increments.
Fecal pH | Fecal samples are collected at three time points: prior to supplementation (earliest 48 hours prior to first visit (day 1)), short after initiation of supplementation (day 3 or soonest thereafter) and again earliest 48 hours prior to last visit (day 15).
  pH of collected fecal samples
Antibody-coating of bacteria | Fecal samples are collected at three time points: prior to supplementation (earliest 48 hours prior to first visit (day 1)), short after initiation of supplementation (day 3 or soonest thereafter) and again earliest 48 hours prior to last visit (day 15).
  Characterization of IgA, IgG and IgM-coating of bacteria from fecal samples using bacterial flow cytometry.
Immunoglobulin G | Results from fasting blood samples taken on day 15 and adjusted for results from day 1 (just before first supplement/placebo dose).
  Plasma immunoglobulin G (g/l)
Immunoglobulin A | Results from blood samples taken on day 15 (just before last supplement/placebo dose) and adjusted for results from day 1 (just before first supplement/placebo dose).
  Plasma immunoglobulin A (g/l)
Leucocyte counts | Results from fasting blood samples taken on day 15 and adjusted for results from day 1 (just before first supplement/placebo dose).
  Total leucocytes as well as basophils, eosinophils, lymphocytes, monocytes, neutrophils as well as the joint group of metamyelo-, myelo- and promyelocytes. All counted in whole blood samples (10^9/l).
Hemoglobin | Results from blood samples taken on day 15 (just before last supplement/placebo dose) and adjusted for results from day 1 (just before first supplement/placebo dose).
  Hemoglobin measured in whole blood (mmol/l).
Alanine transaminase | Results from fasting blood samples taken on day 15 and adjusted for results from day 1 (fasting just before first supplement/placebo dose).
  Plasma alanine transaminase (ALT, U/l) as a biomarker of liver function.
Alkaline phosphatase | Results from blood samples taken on day 15 (just before last supplement/placebo dose) and adjusted for results from day 1 (just before first supplement/placebo dose).
  Alkaline phosphatase (U/l) as a biomarker of liver function.
Aspartate aminotransferase | Results from blood samples taken on day 15 (just before last supplement/placebo dose) and adjusted for results from day 1 (just before first supplement/placebo dose).
  Aspartate aminotransferase also known as aspartate transaminase measured in plasma (U/l) as a biomarker of liver damage.
Bilirubin | Results from blood samples taken on day 15 (just before last supplement/placebo dose) and adjusted for results from day 1 (just before first supplement/placebo dose).
  Bilirubins measured in plasma (µmol/L) as a biomarker of liver function.
Coagulation factors II + VII + X | Results from blood samples taken on day 15 (just before last supplement/placebo dose) and adjusted for results from day 1 (just before first supplement/placebo dose).
  Coagulation factors II + VII + X (INR: International Normalized Ratio) measured in plasma as a biomarker of liver function.
Lactate dehydrogenase (LDH) | Results from blood samples taken on day 15 (just before last supplement/placebo dose) and adjusted for results from day 1 (just before first supplement/placebo dose).
  Lactate dehydrogenase measured in plasma (U/l).
Creatinine | Results from blood samples taken on day 15 (just before last supplement/placebo dose) and adjusted for results from day 1 (just before first supplement/placebo dose)
  Plasma creatinine (µmol/L) as a biomarker of kidney function.
eGFR | Results from blood samples taken on day 15 (just before last supplement/placebo dose) and adjusted for results from day 1 (just before first supplement/placebo dose).
  Estimated glomerular filtration rate (eGFR/ 1,73m² (ml/min)) as a biomarker of kidney function.
Albumin | Results from blood samples taken on day 15 (just before last supplement/placebo dose) and adjusted for results from day 1 (just before first supplement/placebo dose).
  Albumin measured in plasma (g/l).
25-OH-vitamin D | Results from blood samples taken on day 15 (just before last supplement/placebo dose) and adjusted for results from day 1 (just before first supplement/placebo dose).
  Plasma 25-OH-vitamin D (D3+D2) (nmol/L)
TSH | Results from blood samples taken on day 15 (just before last supplement/placebo dose) and adjusted for results from day 1 (just before first supplement/placebo dose).
  Thyroid-stimulating hormone (TSH) measured in plasma (mU/L)
Blood pressure | Measured on day 1 and then again on day 15
  Blood pressure (mm Hg) defined as the lowest value obtained across three measurements.

CONTACTS AND LOCATIONS:
Overall Officials: Jette Frederiksen, Prof, MD, Principal Investigator — Copenhagen University Hospital, Rigshospitalet-Glostrup
Locations (1):
- Optic Neuritis Clinic, Danish Multiple Sclerosis Center, Department of Neurology, Copenhagen University Hospital, Rigshospitalet-Glostrup, Glostrup Municipality, Denmark

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in published articles, after deidentification (text, tables, figures, and appendices).
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: Beginning 3 months and ending 5 years following publication of the article they are presented in.
Access Criteria: Researchers who provide a methodologically sound proposal can access the IPD to achieve the aims of the approved proposal. Proposals should be directed to jette.lautrup.battistini@regionh.dk. To gain access, data requestors will need to sign a data access agreement. Data and explanatory files will be made available at a third party website.

DOCUMENTS (1):
  • Statistical Analysis Plan (2025-07-16): https://cdn.clinicaltrials.gov/large-docs/14/NCT07105514/SAP_000.pdf